CLINICAL TRIAL: NCT05594810
Title: The Feasibility and Potential Efficacy of Adding Tobacco Treatment Using EMDR (ToTEM) to a Regular Smoking Cessation Program A Pilot Randomized Controlled Trail in Inpatient Daily Smokers With a Substance Use Disorder
Brief Title: Tobacco Treatment Using EMDR (ToTEM)
Acronym: ToTEM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too many eligible patients who did not want to participate, very low inclusion rate
Sponsor: IrisZorg (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ToTEM
Record Dates: First submitted 2022-10-07; First posted 2022-10-26 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Tobacco Use Disorder
Keywords: Addiction; Tobacco; EMDR
MeSH Terms: conditions — Tobacco Use Disorder; Behavior, Addictive | interventions — Urocortins

STUDY DESIGN:
Intervention Model Description: Study design: a pilot study with a two-armed randomized controlled design is used in which AF-EMDR + Treatment As Usual (TAU) (Community Reinforcement Approach (CRA) aimed at SUD + a SCP) is contrasted with TAU-only with an intervention phase of three weeks pre- and post intervention assessments and a follow-up after one and three months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU only: Community Reinforcement Approach (CRA) + a regular smoking cessation program (Active Comparator): TAU only
  Interventions: Behavioral: TAU only: Community Reinforcement Approach (CRA) + SCP
- TAU + Addiction focussed - eye movement desensitization and reprocessing (AF-EMDR) + TAU (CRA) (Experimental): TAU + Addiction focussed - eye movement desensitization and reprocessing (AF-EMDR)
  Interventions: Behavioral: TAU + Addiction focussed - eye movement desensitization and reprocessing (AF-EMDR); Behavioral: TAU only: Community Reinforcement Approach (CRA) + SCP

INTERVENTIONS:
Behavioral: TAU + Addiction focussed - eye movement desensitization and reprocessing (AF-EMDR) — A total of six 45-90 min. sessions of AF-EMDR therapy with an average frequency of twice per week added to a SCP embedded in CRA. AF-EMD therapy consists of a rationale, installating a treatment goal, desensitasing mental video's, installation of positive cognition, future template and positive ending.
  Other Names: AF-EMDR
  Arms: TAU + Addiction focussed - eye movement desensitization and reprocessing (AF-EMDR) + TAU (CRA)
Behavioral: TAU only: Community Reinforcement Approach (CRA) + SCP — CRA is a comprehensive cognitive behavioural treatment that focuses on helping people discover and adopt a pleasurable, social and healthy lifestyle that is more rewarding than a lifestyle including substance use.
  Within CRA a regular smoking cessation program is embedded.
  Other Names: CRA (+SCP)

SUMMARY:
Rationale: It is well established that tobacco use has severe health consequences. The prevalence of Tobacco Use Disorder (TUD) is among the highest in populations with Substance Use Disorders (SUD). Despite behavioral and pharmacological treatment options, relapse rates remain high. Therefore, there is a need for additional smoking cessation treatment options that aid long-term abstinence.

A potential interesting intervention is addiction-focused Eye Movement Desensitization and Reprocessing (AF-EMDR) therapy. However, the limited research on AF-EMDR therapy and mixed findings thus far prohibit clinical use. Recently, on the basis of diverse findings thus far, an adjusted AF-EMDR protocol has been developed.

DETAILED DESCRIPTION:
SUMMARY

Rationale: It is well established that tobacco use has severe health consequences. The prevalence of Tobacco Use Disorder (TUD) is among the highest in populations with Substance Use Disorders (SUD). Despite behavioral and pharmacological treatment options, relapse rates remain high. Therefore, there is a need for additional smoking cessation treatment options that aid long-term abstinence.

A potential interesting intervention is addiction-focused Eye Movement Desensitization and Reprocessing (AF-EMDR) therapy. However, the limited research on AF-EMDR therapy and mixed findings thus far prohibit clinical use. Recently, on the basis of diverse findings thus far, an adjusted AF-EMDR protocol has been developed.

Objective: to investigate areas of uncertainty about a possible future definitive RCT using AF-EMDR as an add-on intervention to a Smoking Cessation Program (SCP), by determining:

* Feasibility/process outcomes (e.g. recruitment, adherence, treatment fidelity).
* Preliminary clinical efficacy in order to estimate the effect size for a future power analysis.

Study design: a pilot study with a two-armed randomized controlled design is used in which AF-EMDR + Treatment As Usual (TAU) (Community Reinforcement Approach (CRA) aimed at SUD + a SCP) is contrasted with TAU-only with an intervention phase of three weeks pre- and post intervention assessments and a follow-up after one and three months.

Study population: daily smoking adults, admitted to an inpatient addiction care clinic. A total of 50 eligible participants will be allocated at random to one of two treatment groups.

- In order to be eligible, patients must meet the following criteria: 1) age ≥ 18 years, 2) good Dutch language proficiency, 3) a DSM-5 diagnosis of Tobacco Use Disorder, 4) smoking, on average, ≥ 10 cigarettes per day pre-admission, 5) A score of at least 5 on a scale from 0 to 10, for motivation and self-efficacy, 6) a planned inpatient stay of ≥ 4 weeks, and 7) written informed consent.

Respondents who demonstrate serious therapy interfering behavior or symptoms that also interfere with TAU will be excluded from participation in this study (e. g. psychiatric or medical crisis that requires immediate intervention).

Intervention: a total of six 45-90 min. sessions of AF-EMDR twice per week added to a SCP embedded in TAU.

Main study parameters/endpoints:

* Feasibility, design, recruitment and protocol issues.
* Changes in tobacco craving and smoking behavior.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Tobacco Use Disorder according to the DSM-5 (American Psychiatric Association, 2013) criteria.
* Age ≥ 18 years.
* Good Dutch language proficiency (based on clinical judgement).
* Smoking, on average, ≥ 10 cigarettes per day pre-admission.
* A score of at least 5 on a scale from 0 to 10, for motivation and self-efficacy
* A planned inpatient stay of ≥ 4 weeks.
* Written informed consent.

Exclusion Criteria:

• Serious therapy interfering behavior or symptoms that also interfere with TAU, based on clinical judgement (e. g. psychiatric or medical crisis that requires immediate intervention).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Retention of participants | 1 year
  The retention of participants from randomization until the last follow-up.
Acceptability in terms of compliance | 1 year
  The acceptability of AF-EMDR to participants in terms of compliance, measured by the total number of sessions attended and the proportion of attended versus non attended (planned) sessions; a higher proportion of attended sessions reflects better compliance.
Acceptability in terms of adherence | 1 year
  The acceptability of AF-EMDR to therapists in terms of adherence to the protocol, measured by the score of an independent rater on a self-developed, a-priori established adherence rating protocol using 47 Likert-type items (range 1-5); a higher score reflects better adherence.

SECONDARY OUTCOMES:
Proportion of participants | 1 year
  The proportion of patients at the clinic that are potentially eligible and provide informed consent.
The feasibility of the outcome measures | 1 year
  The feasibility of the outcome measures in terms of completion of questionnaires (% per questionnaire and total).
Missing data | 1 year
  Amount of missing data, measured by total number of missing values and the proportion of completed versus missing data.

OTHER OUTCOMES:
Demographics | 1 year
  Demographics, as inventoried by a structured interview and patient files.
Smoking history | 1 year
  Smoking (cessation history), inventoried by a structured interview and patient files.
DSM-5 | 1 year
  Current DSM-5 diagnoses, inventoried by a structured interview and patient files.
Motivation | 1 year
  Motivation to quit smoking, measured by a Likert-type scale from 0 to 10; a higher score reflects a higher motivation.
Self-efficacy | 1 year
  Smoking cessation self-efficacy, measured by a Likert-type scale from 0 to 10; a higher score reflects a higher self-efficacy.
Nicotine dependence | 1 year
  Severity of nicotine dependence, measured by the Fagerström Test of Nicotine Dependence, providing a score from 0 to 10; a higher score reflects a more severe dependence.
Time to relapse | 1 year
  Time to relapse (from the end of the AF-EMDR intervention, if abstinence is achieved), measured in number of days from the end of the AF-EMDR intervention until first cigarette smoked. The higher the number of days, the longer the time to relapse.
Smoking behavior | 1 year
  Changes from baseline (T0) to T1-T2-T3 in: Smoking behavior, measured by mean number of cigarettes smoked per day over the past 7 days; a higher score means a worse outcome.
Tobacco craving | 1 year
  Changes from baseline (T0) to T1-T2-T3 in: Tobacco craving, as measured by the total score on the Questionnaire of Smoking Urges - Brief version; a higher score means a worse outcome.
Craving related self-control/self-efficacy | 1 year
  Changes from baseline (T0) to T1-T2-T3 in: Craving related self-control/self-efficacy. As measured by a five-item subscale of the Self-control cognitions Questionnaire Likertscales, range 1-5, min 5, max 25); a higher score means a worse outcome.
Positive incentive value | 1 year
  Changes from baseline (T0) to T1-T2-T3 in: Positive incentive value. As measured by a six-item subscale of the Self-control cognitions Questionnaire (Likert-type scales, range 1-5, min. score 6, max 30); a higher score means a worse outcome.
Level of Urge | 1 year
  Within AF-EMDR session changes in: Mean Level of Urge, measured by a Likert-type scale from 0 to 10; a higher score means a worse outcome.
Level of Positive Affect | 1 year
  Within AF-EMDR session changes in: Mean Level of Positive Affect, measured by a Likert-type scale from 0 to 10; a higher score means a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Addiction clinic 'Tiel' IrisZorg, Tiel, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Depending on the final data collection and the journal in which these are published, we will decide on availability of IPD